CLINICAL TRIAL: NCT02050750
Title: Breast Cancer Bank of Tissue From Trial Assigning Individualized Options for Treatment (TAILORx Tissue Bank)
Brief Title: TAILORx Tissue Bank
Status: Active, not recruiting | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 12-30
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Must have registered with the ICORG 06-31 TAILORx trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TAILORx ICORG 06-31: Patients must have participated in TAILORx ICORG 06-31, participated in trial arms, and have adequate tumour tissue available

SUMMARY:
This is an exploratory, translational, non-interventional and multi-centre biobank. The aim of the development of such a biobank is to identify potential biomarkers that are indicative of disease relapse.

DETAILED DESCRIPTION:
The primary objective is to develop a biobank, tissue microarrays (TMAs) and full face sections, which will be used to identify candidate/ novel biomarkers prognostic for disease relapse and predictive for endocrine and/or chemotherapy resistance.

The secondary objectives are:

* To validate emerging signatures/biomarkers identified.
* To develop new assays for the breast cancer clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were registered with the ICORG 06-31 TAILORx trial and participated in trial arms
* Patients with adequate tumor tissue available

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist only of patients that participated in the TAILORx ICORG 06-31 trial. These patients must have participated in trial arms relevant to ICORG 06-31 study and have adequate tumour tissue available.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Disease relapse, endocrine and/or chemotherapy resistance prognosis | For duration of follow up, expected 10 years
  A biobank, TMAs and full face sections, will allow for the identification of candidate/novel biomarkers prognostic for disease relapse and predictive for endocrine and/or chemotherapy resistance

SECONDARY OUTCOMES:
Signature/biomarkers | For the duration of follow up, expected 10 years
  Validation of emerging signature/biomarkers

CONTACTS AND LOCATIONS:
Locations (12):
- Ireland (12):
  - Bons Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Letterkenny General Hospital, Donegal
  - Adelaide and Meath National Children's Hospital Tallaght, Dublin
  - St Vincent Universtiy Hospital, Dublin
  - St James Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Galway University Hospital, Galway
  - Midwestern Regional Hospital, Limerick
  - Sligo General Hosptial, Sligo
  - Waterford Regional Hospital, Waterford

REFERENCES:
- [Derived] Lynch SM, Russell NM, Barron S, Wang CA, Loughman T, Dynoodt P, Fender B, Lopez-Ruiz C, O'Grady A, Sheehan KM, Fay J, Amberger-Murphy V, Saha A, Klinger R, Gonzalez CA, Al-Attar N, Rahman A, O'Leary D, Lanigan FT, Bracken AP, Crown J, Kelly CM, O'Connor DP, Gallagher WM. Prognostic value of the 6-gene OncoMasTR test in hormone receptor-positive HER2-negative early-stage breast cancer: Comparative analysis with standard clinicopathological factors. Eur J Cancer. 2021 Jul;152:78-89. doi: 10.1016/j.ejca.2021.04.016. Epub 2021 Jun 2. PMID 34090143